CLINICAL TRIAL: NCT06056882
Title: Simultaneous CLE Guided Crybiopsy in Patients With Pulmonary Nodules
Status: Recruiting | Type: Observational
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniela Gompelmann, Prof. Dr. med., University of Vienna
Other Study IDs: 1.1
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Other: CLE-guided cryobiopsy

INTERVENTIONS:
Other: CLE-guided cryobiopsy — During bronchoscopy, that is performed for suspicious pulmonary lesions, it is planned to use the CLE probe and cryoprobe simultaneously wafter detection of the round focus.

SUMMARY:
It is planned to use the CLE probe and cryoprobe simultaneously after detection of the round focus.

It is planned to include 5 patients with suspected central airway invading lung carcinoma and 15 patients with suspected peripheral lung carcinoma who have an indication for bronchoscopic histologic confirmation.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Suspicion of lung carcinoma

Exclusion Criteria:

* Known allergy to fluorescin
* Pregnancy and/or lactation
* No discontinuation of ß-blocker 12 hours before intervention possible

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for bronchoscopy and biopsy for suspicious pulmonary lesions
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility | during bronchoscopy procedure
  Advers events

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gompelmann, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No